CLINICAL TRIAL: NCT07219147
Title: Pilot Study of ¹⁷⁷Lu-PSMA-617 in Combination With Sipuleucel-T in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: 177^Lu-PSMA-617 in Combination With Sipuleucel-T for the Treatment of Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25161; NCI-2025-07470 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25161 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-Resistant Prostate Adenocarcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Leukapheresis; Pluvicto; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II; sipuleucel-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (177^Lu-PSMA-617) (Active Comparator): Patients receive 177^Lu-PSMA-617 IV. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, PSMA PET/CT, bone scan, and MRI throughout the study. Additionally, patients may undergo MRI or CT of the brain throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan; Biological: Sipuleucel-T
- Arm B (177^Lu-PSMA-617, sipuleucel-T) (Experimental): Patients receive 177^Lu-PSMA-617 IV. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Starting during week 8 of treatment, patients receive sipuleucel-T IV over 1 hour. Treatment repeat every 2 weeks for up to 3 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo leukapheresis, blood sample collection, PSMA PET/CT, bone scan, and MRI throughout the study. Additionally, patients may undergo MRI or CT of the brain throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Leukapheresis; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan; Biological: Sipuleucel-T

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT and PSMA PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
  Arms: Arm B (177^Lu-PSMA-617, sipuleucel-T)
Drug: Lutetium Lu 177 Vipivotide Tetraxetan — Given IV
  Other Names: 177Lu-labeled PSMA-617; 177Lu-PSMA-617; AAA 617; AAA-617; AAA617; Lu177-PSMA-617; Lutetium Lu 177-PSMA-617; LUTETIUM LU-177 VIPIVOTIDE TETRAXETAN; Lutetium-177-PSMA-617; Pluvicto
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: PSMA PET Scan — Undergo PSMA PET/CT
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography
Biological: Sipuleucel-T — Given IV
  Other Names: APC 8015; APC-8015; APC8015; APC8015 Vaccine; PA2024 (PAP/GM-CSF)-Loaded Dendritic Cell Vaccine; Provenge; SipT

SUMMARY:
This phase I trial compares the effect of lutetium Lu 177 (177^Lu)-prostate-specific membrane antigen (PSMA)-617 in combination with Sipuleucel-T to 177^Lu-PSMA-617 alone in treating patients with prostate that has spread from where it first started (primary site) to other places in the body (metastatic) and has continued to grow and spread despite surgical or medical intervention to block androgen production (castration-resistant). 177^Lu-PSMA-617, a type of radioconjugate, binds to a protein called PSMA, which is found on some prostate tumor cells. It gives off radiation that may kill the tumor cells. Sipuleucel-T, a type of vaccine and a type of cellular adoptive immunotherapy, is made from immune system cells. The cells are treated with a protein that is made by combining a protein found on prostate tumor cells with a growth factor. When the cells are injected back into the patient, they may stimulate T cells to kill prostate tumor cells. Giving 177^Lu-PSMA-617 in combination with sipuleucel-T may be safe, tolerable, and/or effective compared to 177^Lu-PSMA-617 alone in treating patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the immune response induced by the combination of lutetium Lu 177 vipivotide tetraxetan (177^Lu-PSMA-617) and sipuleucel-T, using changes in anti-prostatic acid phosphatase (PAP) immunoglobulin G (IgG) antibody titers.

SECONDARY OBJECTIVES:

I. To evaluate anti-PA2024 antibody titers in patients receiving 177^Lu-PSMA-617 alone versus in combination with sipuleucel-T.

II. To assess the safety and tolerability of 177^Lu-PSMA-617 plus sipuleucel-T. III. To evaluate the clinical efficacy of 177^Lu-PSMA-617 alone versus in combination with sipuleucel-T.

EXPLORATORY OBJECTIVES:

I. To characterize the pharmacokinetics (PK) of 177^Lu-PSMA-617 plus sipuleucel-T in the blood.

II. To determine the impact of 177^Lu-PSMA-617 in combination with sipuleucel-T on systemic immunomodulation.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A (CONTROL GROUP): Patients receive 177^Lu-PSMA-617 intravenously (IV). Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, PSMA positron emission tomography (PET)/computed tomography (CT), bone scan, and magnetic resonance imaging (MRI) throughout the study. Additionally, patients may undergo MRI or CT of the brain throughout the study.

ARM B (EXPERIMENTAL GROUP): Patients receive 177^Lu-PSMA-617 IV. Treatment repeats every 6 weeks for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Starting during week 8 of treatment, patients receive sipuleucel-T IV over 1 hour. Treatment repeat every 2 weeks for up to 3 doses in the absence of disease progression or unacceptable toxicity. Patients also undergo leukapheresis, blood sample collection, PSMA PET/CT, bone scan, and MRI throughout the study. Additionally, patients may undergo MRI or CT of the brain throughout the study.

After completion of study treatment, patients are followed up at 30 days, every 3 months for up to 1 year then every 6 months until progression followed by survival follow until death or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Male
* Progressive castration-resistant metastatic prostate cancer with pathologically confirmed adenocarcinoma of the prostate without small cell features
* Patients must have either:

  * Measurable disease

    * For extranodal (visceral) lesions (e.g. lung, liver, etc.) to be considered measurable, they must be ≥ 10 mm in one dimension, using spiral CT
    * For lymph nodes to be considered measurable (i.e., target or evaluable lesions), they must be ≥ 20 mm in at least one dimension, using spiral CT
  * OR non-measurable disease

    * All other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions
    * Lesions that are considered non-measurable include bone lesions (only). Progression on first generation ADT
* Patients must have been on androgen deprivation therapy with a gonadotrophin releasing hormone (GnRH) analogue, antagonist, or bilateral orchiectomy (i.e., surgical or medical castration) for at least 3 months prior to study entry and maintain castrate levels of serum testosterone < 50 ng/dL throughout study participation unless intolerant
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3 (within 10 days prior to day 1 of protocol therapy)
* White blood cell (WBC) counts > 2500/uL (within 10 days prior to day 1 of protocol therapy)
* Lymphocyte count ≥ 300/uL (within 10 days prior to day 1 of protocol therapy)
* Platelets ≥ 100,000/mm^3 (within 10 days prior to day 1 of protocol therapy)
* Hemoglobin ≥ 9g/dL (within 10 days prior to day 1 of protocol therapy)

  * NOTE: Red blood cell transfusions are not permitted within 14 days of hemoglobin assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (within 10 days prior to day 1 of protocol therapy) (unless has Gilbert's disease, serum bilirubin level ≤ 3 x ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN (within 10 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) ≤ 3.0 x ULN (within 10 days prior to day 1 of protocol therapy)
* Alkaline phosphatase ≤ 3 x ULN (within 10 days prior to day 1 of protocol therapy) (Patients with documented bone metastases, alkaline phosphatase [ALP] ≤ 5 x ULN)
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance of ≥ 50 mL/min per Cockcroft-Gault formula (within 10 days prior to day 1 of protocol therapy)
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN (within 10 days prior to day 1 of protocol therapy)
* If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants (within 10 days prior to day 1 of protocol therapy)
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.3 x ULN (within 10 days prior to day 1 of protocol therapy)
* If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants (within 10 days prior to day 1 of protocol therapy)
* Seronegative for HIV antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR]) (within 10 days prior to day 1 of protocol therapy)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed. OR
  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* For male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception or abstain from heterosexual activity for the course of the study through at least 4 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Any approved or investigational anticancer therapy, including chemotherapy, hormonal therapy (e.g., androgen receptor [AR] antagonists, 5 alpha reductase inhibitor, estrogen), or radiotherapy, within 4 weeks prior to initiation of study treatment

  * Treatment with any of the following medications or interventions within 28 days of registration:

    * External beam radiation therapy or surgery
    * Chrysanthemum morifolium/Ganoderma lucidum/Glycyrrhiza glabra/Isatis indigotica/Panax pseudoginseng/Rabdosia rubescens/Scutellaria baicalensis/Serona repens supplement (PC-SPES) (or PC-SPEC) or saw palmetto
    * Systemic corticosteroids. Use of inhaled, intranasal, and topical steroids is acceptable
    * Megestrol acetate (Megace®), diethyl stilbestrol (DES), or cyproterone acetate
    * Ketoconazole
    * 5-alpha-reductase inhibitors (e.g., finasteride [Proscar®], dutasteride [Avodart®])
    * High dose calcitriol (1,25[OH]2 vitamin [Vit]D) (i.e., > 7.0 ug/week)
* Prior treatment with 177^Lu-PSMA-617 and/or sipuleucel-T
* Radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before first dose of study treatment
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* Treatment with any investigational vaccine within 2 years of registration or treatment with any other investigational product within 28 days of registration
* Patients with acute leukemias, accelerated/blast-phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma
* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases
* Inability to comply with study and follow-up procedures
* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-05 (Estimated); Primary Completion 2028-07-26 (Estimated); Study Completion 2028-07-26 (Estimated)

PRIMARY OUTCOMES:
Anti-prostatic acid phosphatase (PAP) immunoglobulin G (IgG) antibody response rate | Between week 7 and week 19
  Will be defined as the proportion of patients with an IgG titer > 400. Comparisons between study arms will be performed using the Fisher's exact test. Descriptive statistics will be used to summarize the antibody response rates, and Clopper-Pearson exact 95% confidence intervals will be calculated.
Change in anti-PAP IgG antibody titers | Between week 7 and week 19
  Descriptive statistics will be used to summarize antibody titer levels at each time point. Comparisons between study arms will be performed using the Wilcoxon signed-rank test or Student's t-test, as appropriate.

SECONDARY OUTCOMES:
Change in anti-PA2024 antibody titers | Between week 7 and week 19
  Descriptive statistics will be used to summarize antibody titer levels at each time point. Comparisons between study arms will be performed using the Wilcoxon signed-rank test or Student's t-test, as appropriate.
Incidence of adverse events | Up to 30 days after last dose of study treatment
  Comparison of toxicities will be assessed using Common Terminology Criteria for Adverse Events version (v) 5.0 criteria.
Proportion of patients achieving a ≥ 50% reduction in prostate specific antigen (PSA) levels (PSA50 response rate) | At baseline up to 3 years
  The PSA50 response rate will be calculated for each treatment arm as the proportion of patients achieving PSA50 response among all evaluable patients. A Fisher's exact test will be used to compare response rates between arms.
Objective response rate | Up to 3 years
  The association between treatment arm and overall response as per RECIST v 1.1 criteria (response observed versus not observed) will be examined using Fisher's exact test.
Radiographic progression-free survival (rPFS) | From enrollment to progression or death from any cause, assessed up to 3 years
  Will be evaluated using Prostate Cancer Clinical Trial Working Group 3 and RECIST v 1.1 criteria. The median rPFS will be estimated using the Kaplan-Meier method.
Overall survival | From enrollment to death from any cause, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chehrazi-Raffle, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States